CLINICAL TRIAL: NCT02368639
Title: Feasibility of a Modified Positive Airway Pressure Device to Treat Sleep Disordered Breathing
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated due to recruitment slower than anticipated
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIA-156
Record Dates: First submitted 2015-02-08; First posted 2015-02-23 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Sleep Apnea, Obstructive; Obesity Hypoventilation Syndrome
MeSH Terms: conditions — Sleep Apnea, Obstructive; Obesity Hypoventilation Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Positive airway pressure (PAP) device (Experimental): Fisher & Paykel Healthcare PAP Device. Participants will sleep overnight using themodified positive airway pressure device. Their pressures will be titrated by a qualified sleep technician, they will then be optimised during the night.
  Interventions: Device: Fisher & Paykel Healthcare PAP Device

INTERVENTIONS:
Device: Fisher & Paykel Healthcare PAP Device — The device is a modified version of the Fisher & Paykel Icon continuous positive airway pressure (CPAP) device, which is a fully released product in New Zealand.

SUMMARY:
This study will use a modified version of a positive airway pressure device to supply air to the participant, while undergoing supervised polysomnography. Positive airway pressures are typically applied to many patients with hypoventilation, in this study these pressures will be titrated by a qualified sleep technician. During the night these pressures will be altered to optimise comfort.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18+
* Patients diagnosed with obesity hypoventilation syndrome (OHS) and/or obstructive sleep apnea (OSA) by a practicing sleep or respiratory physician, requiring positive airway pressure (PAP) therapy

Exclusion Criteria:

* Recent cardiac or respiratory arrest
* Gastro intestinal bleeding, ileus or recent gastrointestinal surgery
* Coma, decreased level of consciousness or agitation
* Anatomical or subjective difficulty with airway access e.g. facial surgery, trauma, vomiting upper airway obstruction
* Cerebrospinal fluid leak, abnormalities of the cribiform plate or prior history of head trauma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Apnea hypopnea index (AHI) | 8 hours
  The number of apnea and hypopneas will be measured
Peripheral blood oxygen level (SpO2) | 8 hours
  Peripheral blood oxygen level will be measured

CONTACTS AND LOCATIONS:
Locations (1):
- Fisher & Paykel Healthcare Sleep Laboratory, Auckland, New Zealand